CLINICAL TRIAL: NCT00207064
Title: 5-HT2A-receptor Binding: Implications for the Pathophysiology of Schizophrenia and Effects of Treatment With Antipsychotic Drugs
Brief Title: Neurobiological and Neurocognitive Disturbances in First-episode Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Birte Glenthoj (Other)
Collaborators: Rigshospitalet, Denmark (Other); Copenhagen University Hospital, Hvidovre (Other); Glostrup University Hospital, Copenhagen (Other); The Danish Medical Research Council (Other); Copenhagen Hospital Corporation (Other); University of Copenhagen (Other); AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Birte Glenthoj, Professor of Psychopharmacology and Neuropsychiatry, Danish Center for Neuropsychiatric Schizophrenia Research, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: 363055; H-KF-01-078/97 (Other: Ethical Comitee Copenhagen)
Record Dates: First submitted 2005-09-10; First posted 2005-09-21 (Estimated); Last update posted 2011-09-19 (Estimated); Status verified 2011-09

CONDITIONS: Schizophrenia
Keywords: first-episode; altanserin; 5-HT2A receptors; MRI; fMRI; PPI; P300; P50 gating; endophenotypes; vulnerability indicators; quetiapine
MeSH Terms: conditions — Schizophrenia | interventions — Quetiapine Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: quetiapine

INTERVENTIONS:
Drug: quetiapine — flexible doses according to the clinical condition

SUMMARY:
We want to relate disturbances in first-episode schizophrenic patients in serotonin 5-HT2A receptors, brain structure, brain function, and information processing to each other and to psychopathology. Additionally, we want to examine the influence of 5-HT2A receptor blockade on these disturbances. We expect disturbances in the serotonergic system at baseline to correlate with specific structural and functional changes and with disruption in information processing as measured with psychophysiological and neurocognitive methods - and we expect 5-HT2A receptor blockade to reverse some of the functional and cognitive impairments. We do not expect any effect of treatment on brain structure

DETAILED DESCRIPTION:
Patients and matched healthy controls are examined at baseline and again after the patients have been treated for 6 months with a combined 5-HT2A- and dopamine D2- receptor blocker. We have chosen the atypical antipsychotic compound, quetiapine, for the present study since this drug is characterized by a fast koff/low affinity for the dopamine D2 receptors. The purpose of the study is to examine pathophysiological and neuropsychological mechanisms - not treatment effects. We want to characterize neurobiological and functional endophenotypes or vulnerability indicators and to study their stability over time and their relation to treatment and contemporary psychopathology. To the extent that candidate endophenotypes can be characterized as stable and independent of treatment and contemporary psychopathology they will be analysed together with similar findings from previous (identical)cohorts of schizophrenic patients. Specific disturbances will also be related to candidate genes for schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* First-episode schizophrenia. The controls are matched for age, gender and parental socioeconomic status

Exclusion Criteria:

* Previous antipsychotic treatment, mental retardation, organic brain damage, and for the controls a psychiatric diagnosis or first-degree relatives with a psychiatric diagnosis

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2004-04; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
5-HT2A receptor binding and occupancy (PET) | Baseline and after 6 months
Structural MRI | Baseline and after 6 months
Functional MRI | Baseline and after 6 months
Information procession as measured with psychophysiological methods (P300, PPI, P50 gating ect.) | Baseline and after 6 months
An extensive battery of neurocognitive measures | Baseline and after 6 months

SECONDARY OUTCOMES:
PANSS | Baseline and after 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Birte Glenthoj, MD, DMSc., Study Director — Center for Neuropsychiatric Schizophrenia Research, University of Copenhagen, Psychaitric Center Glostrup, Ndr. Ringvej, DK-2600 Glostrup, Denmark
Locations (3):
- Denmark (3):
  - Neurobiology Research Unit, Rigshospitalet, Copenhagen
  - Center for Neuropsychiatric Schizophrenia Research, University of Copenhagen, Psychiatric Center Glostrup, Glostrup Municipality
  - Danish Research Center for Magnetic Resonance Imaging, Hvidovre Hospital, Hvidovre

REFERENCES:
- [Derived] Jessen K, Mandl RCW, Fagerlund B, Bojesen KB, Raghava JM, Obaid HG, Jensen MB, Johansen LB, Nielsen MO, Pantelis C, Rostrup E, Glenthoj BY, Ebdrup BH. Patterns of Cortical Structures and Cognition in Antipsychotic-Naive Patients With First-Episode Schizophrenia: A Partial Least Squares Correlation Analysis. Biol Psychiatry Cogn Neurosci Neuroimaging. 2019 May;4(5):444-453. doi: 10.1016/j.bpsc.2018.09.006. Epub 2018 Sep 25. PMID 30420252
- [Derived] Ebdrup BH, Skimminge A, Rasmussen H, Aggernaes B, Oranje B, Lublin H, Baare W, Glenthoj B. Progressive striatal and hippocampal volume loss in initially antipsychotic-naive, first-episode schizophrenia patients treated with quetiapine: relationship to dose and symptoms. Int J Neuropsychopharmacol. 2011 Feb;14(1):69-82. doi: 10.1017/S1461145710000817. Epub 2010 Aug 12. PMID 20701823
- [Derived] Ebdrup BH, Glenthoj B, Rasmussen H, Aggernaes B, Langkilde AR, Paulson OB, Lublin H, Skimminge A, Baare W. Hippocampal and caudate volume reductions in antipsychotic-naive first-episode schizophrenia. J Psychiatry Neurosci. 2010 Mar;35(2):95-104. doi: 10.1503/jpn.090049. PMID 20184807
- [Derived] Rasmussen H, Erritzoe D, Andersen R, Ebdrup BH, Aggernaes B, Oranje B, Kalbitzer J, Madsen J, Pinborg LH, Baare W, Svarer C, Lublin H, Knudsen GM, Glenthoj B. Decreased frontal serotonin2A receptor binding in antipsychotic-naive patients with first-episode schizophrenia. Arch Gen Psychiatry. 2010 Jan;67(1):9-16. doi: 10.1001/archgenpsychiatry.2009.176. PMID 20048218
- See also: Center for Neuropsychiatric Schizophrenia Research (CNSR) — http://www.cnsr.dk